CLINICAL TRIAL: NCT05197985
Title: A Stepped Wedge Cluster Randomized-control Trial to Improve Child Outcomes Through Caregiving in Cambodia
Brief Title: Improve Child Outcomes Through Caregiving in Cambodia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding cut.
Sponsor: RTI International (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Merseth King, Director, Early Childhood Development, RTI International
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: RTIInternational
Record Dates: First submitted 2021-12-10; First posted 2022-01-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Child Development
Keywords: Cambodia; Nurturing Care; Caregiving; Child Outcomes; ECD

STUDY DESIGN:
Intervention Model Description: Longitudinal, randomized-control trial with stepped-wedge research design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data collectors will not know which families have received treatments. The investigators will be masked during analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Early Childhood Development Intervention (Experimental): Integrated Early Childhood Development Intervention is one intervention package. Inclusion criteria are adults (age 18+) who are primary caregiver of one or more children under the age of 5 years; and pregnant women (age 18+).
  Interventions: Behavioral: IECD Intervention
- Control Arm (No Intervention): This is the control arm that receives no intervention. Inclusion criteria are adults (age 18+) who are primary caregiver of one or more children under the age of 5 years; and pregnant women (age 18+).

INTERVENTIONS:
Behavioral: IECD Intervention — The Nurturing Care curriculum contains: 1) responsive caregiving, 2) the important role everyone plays in raising a child, 3) maternal health and nutrition, 4) responsive feeding and good nutrition, 5) how children grow and develop, 6) hygiene, 7) language development, 8) the importance of play, 9) managing the stress of parenting, 10) protecting your child from harm. Modules will be delivered through group sessions for caregivers, individualized home visits and Social Behavior Change Communication. IECD will build families' capacity to grow and raise healthy food to consume themselves, and connect them to agricultural markets. Specifically, IECD will provide agriculture technical training to Village Model Farms and households, and will facilitate linkages to markets by identifying buyers and connecting them to the farmers. IECD will train and support volunteers to conduct disability screening, and train disability interventionists to provide appropriate therapies and support services.
  Arms: Integrated Early Childhood Development Intervention

SUMMARY:
This study is a longitudinal, randomized-controlled study with a stepped-wedge research design. The Integrated Early Childhood Development Activity (IECD) will implement interventions in three cohorts of villages sequentially across two provinces of Cambodia, Kampong Thom and Preah Vihear. IECD will collect data from all three cohorts together, four times, at 12-month intervals: a baseline prior to any program intervention, a Cohort 1 end line, a Cohort 2 end line and a Cohort 3 end line. IECD's Theory of Change is that by changing caregivers' practices in rearing their children under age 5, those children will demonstrate improvements in child development outcomes. The investigators will use 6 instruments to collect this data, including well-established internationally validated measures. The IECD team enrolled 1,790 households in Preah Vihear and Kampong Thom in June and July 2021. The study will be competed in 2025.

DETAILED DESCRIPTION:
IECD's approach is based on the Nurturing Care Framework, which is a globally adopted conceptual framework for inclusive, integrated early childhood development (ECD). The Nurturing Care Framework describes five indivisible elements of support young children need to thrive: nutrition, health, responsive caregiving, early learning, and protection. IECD addresses these five elements cohesively within the broader ecosystem of families, communities, service providers, and the policy environment to achieve optimal child outcomes (Exhibit 1). Through Objective 1 activities, IECD will create optimal conditions for all children's development by building the skills of families, health providers, and community leaders to provide and promote Nurturing Care. Through Objective 2, IECD will address children's physical development by improving families' abilities to produce or procure nutritious foods; by helping families generate income to support livelihoods; by promoting consumption of nutritious diets; and by strengthening the integration hygiene, health services, and ECD services. Under Objective 3, IECD will leverage existing screening tools to identify children at risk for developmental delays and disabilities, increase referrals, and strengthen local capacity to provide specialized care.

At the end of IECD, more Cambodian children will be thriving and meeting key growth and developmental milestones. Households will have made substantive changes in their behavior in providing responsive caregiving, nutritious diets, and a hygienic environment for young children, as well as in increasing their incomes through market-led agriculture. Caregivers of children with developmental delays and disabilities will have increased access to early identification and quality intervention services. Service providers from across sectors will be actively supporting families of young children with and without disabilities to provide nurturing care. Civil society partners and other stakeholders will have a common understanding of nurturing care priorities and will be aligning their activities in support of improved child outcomes. The ecosystem in which families and service providers interact with each other, with the private sector, and with the Royal Government of Cambodia (RGC) will have shifted toward an enabling environment in which all actors prioritize and operationalize quality, integrated ECD services for all young children.

A. IECD will sustainably change caregivers' practices in Nurturing Care by delivering an IECD Nurturing Care curriculum, which targets caregivers' Key Behaviors with respect to nutrition, health and water sanitation and hygiene (WASH), responsive care and early learning, safety and security, and gender equity in the household. For each of these domains, IECD has identified Key Behaviors of caregivers that when implemented consistently have been shown to improve child outcomes. Messages, examples, modeling and practice are all strategies incorporated into the IECD Nurturing Care curriculum to promote behavior change. This Nurturing Care curriculum will be delivered through:

* Group sessions for caregivers that cover the curriculum in bi-weekly groups (not exceeding 15 people) at the village level, facilitated by Village Health Support Groups (VHSGs), according to session scripts provided by IECD
* Individualized home visits for most vulnerable households, aligned to the same IECD Nurturing Care curriculum, conducted by VHSGs and tailored to the needs of each household
* Cross-cutting Social Behavior Change Communication: mass media and interpersonal communication aimed at changing knowledge, attitudes and practices at the community level to support Nurturing Care.

B. IECD will increase access to healthy and nutritious food by building families' capacity to grow and raise healthy food to consume themselves, and by connecting families to agricultural markets so they can generate income. The specific approaches to achieve these outcomes are:

* Enhanced Homestead Food Production activities, including agriculture technical training to Village Model Farms and households, to ensure all target participants have capacity to increase their agriculture production.
* Linkages to Markets; Field Officers will work with the Nutrition Sensitive Agriculture Coordinator to identify buyers and connect them to the farmers to ensure when the farmers produce agricultural products they could sell out with suitable price.

C. IECD will increase screening for developmental delays and disabilities by scaling up the use of the Cambodian Community-based Developmental Milestone Assessment Tool (Cb-DMAT), and building capacity for therapeutic services for referral of families that need support by:

* Training and supporting VHSGs and other community members to conduct community-based screening
* Training an expanded cadre of disability interventionists to provide appropriate therapies and support services

The study will measure two primary outcomes (development of children aged 6-23 months; and development of children aged 24-59 months), and four secondary outcomes (caregiving practices, women's nutritional status, breastfeeding, children's nutritional status).

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18+) caregivers of one or more child(ren) under the age of 5 years old
* Adult (age 18+) pregnant women

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3500 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
Caregiver Report of Early Development Index (CREDI Instrument) - Child Development | 12 months
  This instrument is used to measure the primary outcome of child development. It is a caregiver-reported questionnaire to measure of developmental status of children aged 6-23 months across developmental domains. The developmental domains are:
  1. Motor Skills (fine and gross)
  2. Language (receptive and expressive)
  3. Cognition (executive function, problem solving & reasoning, and pre-academic knowledge)
  4. Social-Emotional (emotional & behavioral self-regulation, emotional knowledge, social competence)
  5. Mental Health (internalizing, externalizing)
  The scale score is from 0-20. Higher score is optimal. Developed by Harvard. For more information, see https://sites.sph.harvard.edu/credi/.
Early Childhood Development Indicators (ECDI Instrument) - Child Development | 12 months
  This instrument is used to measure the primary outcome of child development. It is a caregiver-reported questionnaire to measure of developmental status of children aged 24-59 months across domains of learning, psychological well-being, and health, and 12 sub-domains. The scale score is from 0-20. Higher score is optimal. Developed by UNICEF. For more information, see https://data.unicef.org/resources/early-childhood-development-index-2030-ecdi2030/.

SECONDARY OUTCOMES:
Integrated Early Childhood Development Caregiving Key Behaviors (ECDI Instrument) | 12 months
  This instrument is used to measure the secondary outcome of caregiving practices. It is a caregiver-reported questionnaire to measure study participants practicing targeted integrated early childhood development key behaviors in ten domains: 1) caregiving interactions; 2) abuse and neglect; 3) facilitating play; 4) communication; 5) responsive feeding; 6) task sharing; 7) gender attitudes; 8) caregiving routine; 9) social safety net; 10) caring for sick child. There are 38 items, based on the United Nations Children's Fund (UNICEF) Nurturing Care framework (for more information, see https://nurturing-care.org/.) The scale score is from 0-38. High score is optimal. Developed by RTI International.
World Health Organization Minimum Acceptable Diet Instrument (children aged 6-23 months) | 12 months
  This instrument is used to measure the secondary outcome of children's nutritional status. It is a caregiver-reported questionnaire which measures the degree to which participating children aged 6-23 months are consuming the minimum acceptable diet, as defined by the World Health Organization. The structure of the questionnaire is a 24-hour dietary recall. Caregivers indicate which items from a list of 8 food groups the child has consumed in the past 24-hours. Scale score from 0-8. High score is optimal.
  For more information, see: https://www.who.int/data/nutrition/nlis/info/infant-and-young-child-feeding.
WHO Prevalence of Exclusive Breastfeeding Instrument (children aged 0-6 months) | 12 months
  This instrument is used to measure the secondary outcome of exclusive breastfeeding of children aged 0-6 months. This is a caregiver-reported questionnaire that collects data on the breastfeeding practices of children participating in the study. The questionnaire include 5 items which cover initiation of breastfeeding, duration of breastfeeding, and exclusivity of breastfeeding. The scale score is from 0-5. High score is optimal.
  For more information, see: http://whqlibdoc.who.int/publications/2010/9789241599290_eng.pdf.
WHO Minimum Dietary Diversity-Women (MDD-W) Instrument | 12 months
  This instrument is used to measure the secondary outcome of women's nutritional status. The instrument is a caregiver-reported questionnaire which measures the degree to which women of reproductive age are consuming a diet of minimum acceptable diversity, as defined by the World Health Organization. The questionnaire is a 24-hour dietary recall, capturing which of ten food groups respondents have consumed in the past day, e.g., dairy, vegetables, animal-source proteins. The scale score is 0-26. High score is optimal.
  For more information, see: https://inddex.nutrition.tufts.edu/data4diets/indicator/minimum-dietary-diversity-women-mdd-w

CONTACTS AND LOCATIONS:
Locations (1):
- RTI International, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Derived] King KM, Yeng S, Brennan C, Creel D, Ames JW, Cotes G, Bann CM, Black MM. Integrated Early Childhood Development in Cambodia: Protocol of a Cluster Stepped-Wedge Trial. Pediatrics. 2023 May 1;151(Suppl 2):e2023060221N. doi: 10.1542/peds.2023-060221N. PMID 37125891